CLINICAL TRIAL: NCT00008242
Title: A Phase II Clinical Trial Of Thalidomide, Adramycin And Dexamethasone (TAD) As Initial Therapy For The Treatment Of Multiple Myeloma
Brief Title: Thalidomide, Doxorubicin, and Dexamethasone in Treating Patients With Untreated Stage II or Stage III Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 00-077; P30CA008748 (NIH); MSKCC-00077; NCI-G00-1893
Record Dates: First submitted 2001-01-06; First posted 2004-05-04 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Dexamethasone; Doxorubicin; Thalidomide

INTERVENTIONS:
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: thalidomide

SUMMARY:
RATIONALE: Thalidomide may stop the growth of multiple myeloma by stopping blood flow to the cancer cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining thalidomide with chemotherapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of thalidomide, doxorubicin, and dexamethasone in treating patients who have untreated stage II or stage III multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate of patients with previously untreated stage II or III multiple myeloma treated with thalidomide, doxorubicin, and dexamethasone. II. Determine the safety and toxicity of this regimen in this patient population.

OUTLINE: Patients receive oral dexamethasone on days 1-4, 9-12, and 17-20, doxorubicin IV on day 1, and oral thalidomide daily. Treatment repeats every 30 days for 4 courses in the absence of unacceptable toxicity or disease progression.

PROJECTED ACCRUAL: A total of 21-45 patients will be accrued for this study within approximately 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed multiple myeloma Stage II disease Symptomatic due to progressive disease OR Stage III disease No stage I multiple myeloma or smoldering myeloma

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-3 Life expectancy: More than 4 months Hematopoietic: Absolute granulocyte count at least 1,500/mm3* Platelet count at least 100,000/mm3* *Unless due to multiple myeloma Hepatic: Bilirubin no greater than 2.0 mg/dL ALT and AST no greater than 3 times upper limit of normal (ULN) Alkaline phosphatase no greater than 3 times ULN Renal: Elevated creatinine allowed Cardiovascular: LVEF at least 50% by MUGA or ECHO No active angina No myocardial infarction within the past 6 months Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception at least 4 weeks prior to, during, and for at least 4 weeks after study No grade II or greater pre-existing neuropathy No other concurrent or prior active malignancy within the past 2 years except adequately treated non-melanoma skin cancer or carcinoma in situ of the cervix Prior T1a or T1b prostate cancer (detected incidentally at transurethral resection of prostate (TURP) and comprising less than 5% of resected tissue) allowed if PSA normal since TURP HIV negative No AIDS-related illness No other medical condition that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for multiple myeloma Endocrine therapy: No more than 1 course of prior pulse dexamethasone Prior steroids of less than 1 month duration for emergent indications or life-threatening lesions (e.g., hypercalcemia or spinal cord compromise) allowed Radiotherapy: Prior radiotherapy allowed Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond L. Comenzo, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Hassoun H, Reich L, Klimek VM, Dhodapkar M, Cohen A, Kewalramani T, Zimman R, Drake L, Riedel ER, Hedvat CV, Teruya-Feldstein J, Filippa DA, Fleisher M, Nimer SD, Comenzo RL. Doxorubicin and dexamethasone followed by thalidomide and dexamethasone is an effective well tolerated initial therapy for multiple myeloma. Br J Haematol. 2006 Jan;132(2):155-61. doi: 10.1111/j.1365-2141.2005.05848.x. PMID 16398649